CLINICAL TRIAL: NCT04859842
Title: Comparison of Effectiveness of Pulsed Electromagnetic Field Therapy and Interferential Current on Patients With Chronic Low Back Pain
Brief Title: Comparison of Two Electrotherapy Methods on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-RK-06
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain, Mechanical
Keywords: Rehabilitation; Electric Stimulation Therapy; Quality of Life; Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Electric Stimulation Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Conventional therapy group will receive sham electrotherapy sessions and outcome assessments will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulse Electromagnetic Field Group (Active Comparator): Pulse Electromagnetic Field Therapy (PEMF) will be applied to patients' low back region. Also, patients will receive a conventional therapy program consisting of hotpack, ultrasound, and transcutaneous electrical stimulation in addition to PEMF therapy.
  Interventions: Other: Pulse Electromagnetic Field
- Interferential Current Group (Active Comparator): Interferential current will be applied to patients' low back pain region. Also, patients will receive a conventional therapy program consisting of hotpack, ultrasound, and transcutaneous electrical stimulation in addition to Interferential current.
  Interventions: Other: Interferential Current
- Sham Group (Sham Comparator): Sham electrodes will be placed on the low back region. Also, patients will receive a conventional therapy program consisting of hotpack, ultrasound, and transcutaneous electrical stimulation in addition to sham therapy.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Pulse Electromagnetic Field — Patients will be treated for two weeks, five days a week, one session a day, and 10 sessions with PEMF in prone position. Each session will be 45 minute long with a 15 minute PEMF therapy and a 30 minute conventional therapy program.
  Arms: Pulse Electromagnetic Field Group
Other: Interferential Current — Patients will be treated for two weeks, five days a week, one session a day, and 10 sessions with Interferential current in prone position. Four interferential electrode will be placed on low back region. Each session will be 45 minute long with a 15 minute interferential current and a 30 minute conventional therapy program.
  Arms: Interferential Current Group
Other: Sham — Patients will be treated for two weeks, five days a week, one session a day, and 10 sessions with conventional therapy and sham electrotherapy. Sham application will be performed on prone position with four electrodes and electrodes will stay for 15 minutes on this region.
  Arms: Sham Group

SUMMARY:
The purpose of this study is; to compare the effects of interferential current therapy (IF) applied in addition to conventional physical therapy on pain, functional status and quality of life compared to pulsed electromagnetic field therapy (PEMF) in patients with chronic low back pain.

DETAILED DESCRIPTION:
The low back is the most common region for musculoskeletal pain. Many factors play a role in the etiology of low back pain. A certain etiological factor or pathophysiological mechanism cannot be found in 85-90% of the patients.

Approximately 80% of those living in industrialized countries experience low back pain in some part of their lives. 10% of low back pain becomes chronic. It is believed that 1% of workforce losses are due to low back pain. This type of pain often occurs when the back muscles, tendons and ligaments are exposed to stress or strain. Mechanical back pains are chronic pain that often affects the lower part of the spine and radiates to the gluteal region. Since daily activities such as leaning, turning, lifting, standing and sitting for a long time increase the pain, the intensity of the pain increases during the day.

Interferential current (IF) therapy is obtained from two medium frequency currents and is applied by delivering a low frequency current (for example 20 to 100 Hz) to the tissue.

Pulsed ElectroMagnetic Field (PEMF) therapy, which is among physical therapy methods, is frequently used in the treatment of knee, hip and spine osteoarthritis symptoms. It is thought that magnetic field therapy improves the oxygen utilization of the cells and the erythrocytes release more oxygen under the influence of the magnetic field, thus having a positive effect on the circulatory system

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with nonspecific low back pain
* Symptom onset with more than 3 months

Exclusion Criteria:

* History of surgery on low back region
* Structural deformity on the low back region
* Radiculopathy
* Tumor or malignancy
* Any skin condition that prevents usage of electrotherapy
* Having a pace maker or other types of implants on the low back, pelvis and thoracic region

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | two weeks
  It contains 11 digits that should be assigned according to the perceived pain intensity on a numerical scale. The participant chooses the number that best reflects his or her pain. In our study, the patients were informed that the '0' point was not pain at all, and the '10' point expressed unbearable pain.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire | two weeks
  It is a questionnaire developed to evaluate functional disabilities in patients with low back pain. Turkish validity and reliability study was conducted in 2001 (20). In the 24-sentence questionnaire about functional impairments, patients are asked to answer each sentence as yes if it fits their situation, and no if it does not. Yes responses are calculated as "1" and no answers are calculated as "0" points. In this questionnaire with a total score between 0-24, the higher score means more disability.
Euroqol Quality Of Life Scale | two weeks
  EQ-5D is a self-report scale developed by the EuroQoL group, the Western European quality of life research community, and evaluates five dimensions with 1 question each. These five dimensions consist of subtitles of mobility, self-care, usual daily activities, pain / discomfort and anxiety / depression. The answers given to each dimension have 3 options: no problem, some problem and major problem. As a result, 243 possible different health outcomes are defined with the scale. An index score ranging from -0.59 to 1 is calculated from the 5 dimensions of the scale. In the score function, a value of 0 indicates death, a value of 1 indicates perfect health, while negative values indicate unconsciousness, living dependent on bed, etc. show situations. Also included in the scale is a VAS (EQ-VAS) that includes answers between 0 and 100, ie "0 = the worst health condition imaginable" and "100 = the best health condition imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University; Ramazan KURUL, Ph.D, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (1):
- Faculty of Health Sciences Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)